CLINICAL TRIAL: NCT04644601
Title: Translation, Cross-cultural Adaptation and and Psychometric Properties of "The Cumberland Ankle Instability Tool (CAIT)" in Italian Language
Brief Title: Italian Version of The Cumberland Ankle Instability Tool (CAIT)
Acronym: CAIT-I
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Angela Contri, Principal Investigator, University of Bologna
Other Study IDs: 273082
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Instability, Joint; Ankle Sprains; Ankle Injuries; Sport Injury; Chronic Instability of Joint; Chronic Instability, Capsular Ligament; Ankle Inversion Sprain
Keywords: Instability; Ankle; Sprain, Translation, Runners
MeSH Terms: conditions — Joint Instability; Ankle Injuries; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Design: Evaluation of the psychometric properties of a translated, culturally adapted questionnaire.

Objective: Translating, culturally adapting, and validating the Italian version of the Cumberland Ankle Instability Tool (CAIT-I), allowing its use with Italian-speaking population to monitor both state of health and functional limitation deriving from ankle instability problems, in order to evaluate the degree of severity, without using the comparison with the opposite limb.

Summary of Background Data: Lateral ankle sprain is the most common injury during sports activity, often cause of disability and of numerous complications following repeated episodes, including chronic ankle instability (CAI), which affects 32% to 74% of the aforementioned cases.

Growing attention is devoted to standardized outcome measures to improve interventions for injured population.

A translated form of the Cumberland Ankle Instability Tool (CAIT), a simple and specific tool for diagnosing chronic lateral ankle instability with excellent psychometric characteristics of both reliability and validity, has never been validated within the Italian speaking population.

DETAILED DESCRIPTION:
The Cumberland Ankle Instability Tool (CAIT) is a simple 9-item, validated and specific tool for diagnosing chronic lateral ankle instability. This rating scale was first published in 2006, and it is a useful tool as a diagnostic criterion, as a screening tool, a prognostic tool, a outcome and clinical picture severity measure tool.

The CAIT-I questionnaire will be developed involving forward-backward translation, a final re-evaluation made by a representative multidisciplinary expert committee and the realization of a prefinal version to establish a proper correspondence with the original English version.

Once an acceptability analysis has been conducted, the following will be analyzed: 1- The validity of the construct by comparing the CAIT-I data with those of the SF-36 using Pearson's correlations ; 2- An Exploratory Factorial Analysis and one of Internal Consistency; 3 Sensitivity analysis through the development of ROC curves and analysis of the area under the curve. In a subset of at least 36 participants the investigators will determine the internal responsiveness on 4 points using an ANOVA (P <.05). The scores of participants with Chronic Instability will be analyzed to determine the presence of ceiling or floor effects. Standard psychometric techniques will be used.

The validation of the psychometric properties of the instrument will start after it will been administered digitally, via a link to a website built using LimeSurvey, an application based on a MySQL database that allows the realization of online surveys, to a sample population of at least 197 subjects (a priori sample number calculated through the G * Power program) aged 18 or more recruited through sports associations and health professionals who work with sports subjects. Through this link, from the time it will be online up to 16 November 2021, the participants will be able to access the online questionnaire, only after accepting a form for requesting consent to the processing of personal data updated pursuant to article 13 of the GDPR 2016 / 679, in force in all European Union countries from 25 May 2018. Inclusion criteria: - Age ≥18 years - Agreement to voluntarily sign informed consent to participate in the study. Exclusion criteria: - Inability to understand the written Italian language - Pregnancy - Having undergone an ankle-foot surgery in the last 6 months.

Upon enrollment, participants will answer a demographics questionnaire, the CAIT-I, and the SF-36. If they will take part in the reliability portion, then they filled out the CAIT-I and SF-36 a second time within 4 to 9 days.

For the statistical analysis standard psychometric techniques will be used, such as reliability assessments, convergent and discriminant validity tests of each item and of the construct in its entirety, empirical validity tests in relation to the clinical status and formal tests to assess their accuracy to ends to test the hypotheses.

The investigators hypothesize to be able to reproduce a tool that reflects the characteristics of the CAIT in the original language and therefore it will prove to have, even in its Italian version, an acceptable psychometric performance as an outcome and screening measure for chronic ankle instability. The CAIT-I will show to be a useful tool that can be used as a functional outcome measure for the Italian population, to monitor both the state of health and residual functional limitation in adults.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Agreement to voluntarily sign informed consent to participate in the study.

Exclusion Criteria:

* Inability to understand the written Italian language
* Pregnancy
* Having undergone a surgery on the ankle-foot area in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects will be invited to partecipate in this study through contacts with the authors and other colleagues.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
CAIT Score | November 2021
  The Cumberland Ankle Instability Tool is a 9-item questionnaire designed to evaluate both ankles concerning pain in each ankle for daily activities, ankle instability in different types of physical activities, ankle control when recurrent sprain occurring and recovery period after recurrent ankle sprains. The nine items generate a total score from 0 to 30 for each foot, in which 0 is the worst possible score, meaning severe instability, 30 is the best possible score, meaning normal stability
Validate the Italian translation of the CAIT-I | November 2021
  The score between the CAIT-I versus the italian validated version of the Short Form Health Survey (SF-36) will be compared

SECONDARY OUTCOMES:
CAIT-I test-retest reliability | November 2021
  Assess CAIT-I test-retest reliability in adults with and without chronic ankle instability. Test-retest reliability will be assessed with 1 group (including "healthy" and "injured" participants), 2 measurements (test-retest), with an effect size change of 0.25, power of 0.95, and a significance level of α = .05. Test-retest reliability analysis separately will compare combined, healthy, and injured groups for the CAIT total score. The ICC values of 0.49 or less will be considered low, 0.50 to 0.69 moderate, 0.70 to 0.89 high, and 0.90 to 1.00 very high.
CAIT-I construct validity | June 2022
  Assess CAIT-I construct validity in with 1 group (adult with and without chronic ankle instability), with an effect-size change of 0.25, power of 0.95, and a significance level of α = .05
CAIT-I factor analysis and internal consistency | June 2022
  Assess CAIT-I factor analysis and internal consistency in adults with and without chronic ankle instability. Cronbach's alpha will be calculate to estimate internal item consistency.
CAIT-I sensitivity | June 2022
  Assess CAIT-I sensitivity in adults with and without chronic ankle instability. To conduct sensitivity analyses in the healthy group and injured group, the researchers will conduct a t test for equal variances not assumed and a significant Levene's test.
CAIT-I Internal responsiveness | June 2022
  To determine internal responsiveness, differences in CAIT-I and SF-36 scores in injured participants across 4 time points using repeated-measures (time) analysis of variance in SPSS.
CAIT-I Floor and Ceiling Effects | June 2022
  Assess CAIT-I Floor and Ceiling Effects in the injured group

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Ballardin, BSc, OMPT, Principal Investigator — University of Bologna; Angela Contri, MA, OMPT, Principal Investigator — University of Bologna; Matteo Gaucci, MSc, OMPT, Principal Investigator — University of Bologna; Gian Luca De Marco, BSc, OMPT, Principal Investigator — University of Bologna; Veronica Zannoni, BSc, OMPT, Principal Investigator — University of Bologna
Locations (1):
- Unità Operativa di Medicina del Lavoro AOU Sant'Orsola-Malpighi, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Yes
On request the investigators can provide participants (anonymous) data
Supporting Information: Study Protocol
Time Frame: Forever
Access Criteria: Free

REFERENCES:
- [Background] Harriss DJ, Macsween A, Atkinson G. Standards for Ethics in Sport and Exercise Science Research: 2018 Update. Int J Sports Med. 2017 Dec;38(14):1126-1131. doi: 10.1055/s-0043-124001. Epub 2017 Dec 19. No abstract available. PMID 29258155
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Result] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Result] Wright CJ, Arnold BL, Ross SE, Linens SW. Recalibration and validation of the Cumberland Ankle Instability Tool cutoff score for individuals with chronic ankle instability. Arch Phys Med Rehabil. 2014 Oct;95(10):1853-9. doi: 10.1016/j.apmr.2014.04.017. Epub 2014 May 9. PMID 24814563
- [Result] Gribble PA, Delahunt E, Bleakley C, Caulfield B, Docherty C, Fourchet F, Fong DT, Hertel J, Hiller C, Kaminski T, McKeon P, Refshauge K, van der Wees P, Vicenzino B, Wikstrom E. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. Br J Sports Med. 2014 Jul;48(13):1014-8. doi: 10.1136/bjsports-2013-093175. Epub 2013 Nov 19. PMID 24255768